CLINICAL TRIAL: NCT03034174
Title: Pharmacokinetics of High-dose Tigecycline in Critically Ill Patients: an Observational, Prospective Study
Brief Title: Pharmacokinetics of High-dose Tigecycline in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Medical University of Lublin (Other)
Responsible Party: Principal Investigator, Michał Borys, associate professor, Medical University of Lublin
Other Study IDs: KE-0254/258/2014
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Septic Shock; Antibiotic Resistant Infection; Critical Illness
Keywords: tigecycline; pharmacokinetics
MeSH Terms: conditions — Shock, Septic; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients' arterial blood samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- tigecycline: Each patient will receive: tigecycline (200 mg q 12 hours i.v.), meropenem (2 g q 8 hours i.v). In each case CVVHD will be started.
  Blood samples (3 mL) will be collected 2, 4, 8 and 12 hours after each dose of tigecycline for 3 consecutive days.

SUMMARY:
The objective of this study is to describe the pharmacokinetics of tigecycline in critically ill patients receiving continuous venovenous haemodialysis (CVVHD) and to evaluate the frequency of pharmacokinetic/pharmacodynamic target attainment with high dosing strategy (200 mg loading dose and 100 mg/12h).

DETAILED DESCRIPTION:
This is a prospective observational study performed on critically ill patients. Inclusion criteria are: severe sepsis on admission requiring broad-spectrum antibiotics. Both medical and surgical patients will be included. Any type of infections will be included (pulmonary, abdominal, urinary tract, etc.) Antibiotics regimen includes: tigecycline (200 mg every 12 hours intravenously), meropenem (2 grams every 8 hours intravenously).

Blood samples (3 mL) will be collected 2, 4, 8 and 12 hours after each dose of tigecycline for 3 consecutive days. The standard arterial canula will be used to obtain samples.

In each case CVVHD will be started and continued for at least 3 days' period. 30 minutes after a collection each sample will be centrifuged for 10 minutes at 3,000 rpms. Subsequently, supernatant will be collected and frozen.

Serum tigecycline concentration will be measured with high performance liquid chromatography.

Each patient's hemodynamics parameters will be recorded with the use of transpulmonary thermodilution technique (PICCO). Other therapies i.e.: ventilatory support, sedation, an antifungal agent will be given as required.

ELIGIBILITY:
Inclusion Criteria:

* Patients who require ICU treatment due to severe sepsis
* age 18-80 years
* CVVHD treatment
* an eligible consent obtained from the patient or his/her attendant

Exclusion Criteria:

* allergy to tigecycline or meropenem
* contraindication to CVVHD
* lack of consent to participate in the study
* age of patients below 18 or above 80 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to ICU due to severer sepsis recognition. Both medical and surgical patients will be included. Any site of infection will be treated in the manner.
  In each case CVVHD will be initiated and continued. Each patient will receive 200 mg tigecycline q 12h, 2 g meropenem q 8 h. Other treatment as required.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Serum concentration of tigecycline | 72 hours for each patient from the tigecycline treatment initiation.
  Samples obtain from ICU patients 2, 4, 8 12 hours after each dose of tigecycline for 3 days.

CONTACTS AND LOCATIONS:
Overall Officials: Mirosław Czuczwar, M.D. PhD., Principal Investigator — Medical University of Lublin
Locations (1):
- II Department of Anesthesia and Intensive Care, Medical University of Lublin, Lublin, Poland

IPD SHARING:
Plan to Share IPD: No